CLINICAL TRIAL: NCT02247622
Title: Primary Sclerosing Cholangitis Telomere Length
Brief Title: Telomere Length and Other Parameters of Telomere Dysfunction in PSC and Colitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, ido laish, Md., Meir Medical Center
Other Study IDs: 1.1
Record Dates: First submitted 2013-07-10; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Primary Sclerosing Cholangitis; Inflammatory Bowel Disease
Keywords: telomeres; PSC
MeSH Terms: conditions — Cholangitis, Sclerosing; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy control
- IBD: patients with inflammatory bowel disease, study group
- PSC: patients with primary sclerosing cholangitis, study group

SUMMARY:
PSC is a chronic cholestatic disorder. The investigators intend to study some telomere parameters and telomere length in order to predict a premalignant state.

DETAILED DESCRIPTION:
Primary sclerosing cholangitis (PSC) and colitis are chronic inflammatory disorders with malignant potential. Telomerase is an enzyme complex that lengthens telomeres and has enhanced expression in numerous malignancies. In this study, we evaluated the telomerase gene copy number, telomere length, cells in senescence, aneuploidy and additional parameters of telomere dysfunction from peripheral blood lymphocytes of patients.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* documented PSC and inflammatory bowel disease

Exclusion Criteria:

* under 18 years, above 80 y
* known active malignancy
* decompensated cirrhosis
* patients who cannot sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with primary sclerosing cholangitis and inflammatory bowel disease
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Telomere length | 1.5 years

SECONDARY OUTCOMES:
number of cells with increased telomerase RNA component (TERC) expression | 1.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Derived] Laish I, Katz H, Stein A, Liberman M, Naftali T, Kitay-Cohen Y, Biron-Shental T, Konikoff FM, Amiel A. Telomere dysfunction in peripheral blood lymphocytes from patients with primary sclerosing cholangitis and inflammatory bowel disease. Dig Liver Dis. 2015 Sep;47(9):790-6. doi: 10.1016/j.dld.2015.05.002. Epub 2015 May 13. PMID 26048252